CLINICAL TRIAL: NCT06253637
Title: Daratumumab in Very High-Risk T-Lineage Acute Lymphoblastic Leukemia (ALL) Treated According to the ALL National Treatment Program (DARATALL-VHR)
Brief Title: Daratumumab in VHR T-ALL Treated According to the ALL National Treatment Program
Acronym: DARATALL-VHR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALL3024
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: T-Lymphocytic Leukemia, Acute
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Very high risk T-ALL patients treated with daratumumab and the national treatment program (Experimental): After a steroid/cyclophosphamide pre-treatment phase, patients will be treated according to the national treatmetn program - as per the previous GIMEMA LAL1913 - plus daratumumab as follows:
  * In the first cycle, C1, daratumumab (subcutaneous) 1800 mg will be administered on days 1, 8, 15 and 22
  * In the second cycle, C2, daratumumab 1800 mg will be administered on days 1, 8, 15
  * In the subsequent cycles C3-C8 daratumumab 1800 mg will be administered on day 1
  in addition to chemotherapy according to the national treatment program
  Induction/consolidation cycles are administered at 28 (C1-2) and 21(C2-8) day intervals. Dose reductions are required in patients > 55y
  All patients are eligible for allo-SCT after C3. All patients unable to undergo an allo-SCT are eligible for an auto-SCT after C8, If unable to undergo an auto-SCT, these patients are eligible to maintenance at the end of the consolidation program.
  Interventions: Drug: Daratumumab plus chemotherapy according to the national treatment program

INTERVENTIONS:
Drug: Daratumumab plus chemotherapy according to the national treatment program — Daratumumab is a human IgG1қ monoclonal antibody that binds with high affinity to a unique epitope on CD38, a transmembrane glycoprotein which is expressed in several hematological malignancies including multiple myeloma (MM) and ALL. Daratumumab induces lysis of CD38-expressing tumor cells by several mechanisms. Intravenous daratumumab has been approved first as a single agent and then in combinations in the MM setting and in AL amyloidosis.
  The activity of daratumumab in ALL is being explored in the DELPHINUS trial, in which the drug was combined with chemotherapy in pediatric and young adult patients with relapsed/refractory T-cell ALL or lymphoblastic lymphoma (LL).
  In the present trial, daratumumab will be administered to adult Very high risk T-lineage ALL weekly in induction and early consolidation (C1-C2), and the first day of each of the following intensive cycles up to C8.

SUMMARY:
The goal of this clinical trial is to test daratumumab in adult very high risk T-lineage lymphoblastic leukemia.

The main question it aims to answer is wether the addition of daratumumab daratumumab to the national standard of care is able to increase the rate of MRD-negative patients after induction therapy.

Participants will be treated with:

• daratumumab in combination with a pediatric-inspired treatment scheme - as in the previous GIMEMA LAL1913 protocol.

DETAILED DESCRIPTION:
This study is a multicenter phase II trial based on the addition of daratumumab to chemotherapy in the front-line treatment of very high-risk T-ALL.

T-ALL patients are eligible at diagnosis in case of ETP or near ETP immunophenotype. Due to their biological and clinical similarities, T-Myeloid MPAL can also be included. Other VHR T-ALL patients (i.e. those with WBC count >100 x109/L, with complex karyotype with ≥5 unrelated anomalies or with a CD1a-negative immunophenotype) will also be eligible.

A safety run-in is foreseen for 5 patients: if grade >3 infusion-related reactions or extra hematologic adverse events of grade >3 that, for investigator's clinical judgement cannot be due to chemotherapy alone, are not observed in more than 2 patients during the first cycle of daratumumab, the study will continue with the core phase.

After a steroid/cyclophosphamide pre-treatment phase, that can occur before enrollment during the screening period, patients who meet the eligibility criteria will be treated with daratumumab in combination with a pediatric-inspired treatment scheme - as in the previous GIMEMA LAL1913 protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. A diagnosis of T-ALL according to the 2022 International Consensus Classification (ICC) is required, either de novo or secondary to chemo-radiotherapy for another cancer. Pre-treatment with low-dose corticosteroids +/- cyclophosphamide in patients presenting with hyperleukocytosis is allowed.
3. Availability of fresh bone marrow (BM) (or peripheral blood (PB) in patients with hyperleukocytosis) samples to perform diagnostic procedures. ).
4. Bone marrow blast percentage at diagnosis ≥20%.
5. CD38 positivity on ALL blasts (any level of positivity).
6. ETP and near ETP at diagnosis according to internationally accepted criteria (appendix G) at diagnosis or other VHR T-ALL subtypes (WBC count >100 x109/L; complex karyotype with ≥5 unrelated anomalies; other CD1a-negative immunophenotypes). T-Myeloid MPAL according to the 2022 ICC of Acute Leukemias of Ambiguous Lineage (appendix H) can also be eligible and considered as VHR.
7. Availability of full cytological, cytochemical, immunophenotypic, cytogenetic and molecular disease characterization according to the EGIL and WHO classifications.
8. An ECOG performance status 0-2, unless a performance of 3 is unequivocally caused by the disease itself, (and not by pre-existing comorbidities,) and is considered and/or documented to be reversible following the application of anti-leukemic therapy and appropriate supportive measures.
9. For females of childbearing potential, a negative pregnancy test must be documented. Female and male patients who are fertile must agree to use an effective form of contraception with their sexual partners from enrollment through 12 months after the end of treatment.
10. Signed written informed consent according to ICH/E U/GCP and national local laws.

Exclusion Criteria:

1. Diagnosis of B-lineage ALL, and Ph+ ALL.
2. Down's syndrome.
3. Prior systemic chemotherapy for ALL (excluding cyclophosphamide during pre-phase).
4. Pre-existing, uncontrolled pathology such as heart failure (congestive/ischemic, acute myocardial infarction within the past 3 months, untreatable arrhythmias, NYHA classes III and IV), severe liver disease with serum direct bilirubin >3 mg/dL (unless attributable to Gilbert' syndrome or ALL) and/or ALT >5x upper normal limit (unless attributable to ALL), kidney function impairment with serum creatinine >2 mg/dL (unless attributable to ALL), and severe neuropsychiatric disorder that impairs the patient's ability to understand and sign the informed consent, or to cope with the intended treatment plan. N.B. For altered liver and kidney function tests, eligibility criteria can be reassessed at 24-96 hours, following the institution of adequate supportive measures.
5. Presence of serious, active, uncontrolled infections.
6. A history of cancer that is not in a remission phase following surgery and/or radiotherapy and/or chemotherapy, with a life expectancy <2 years.
7. Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
MRD-negativity rate after cycle 1 | 1 month
  Number of patients on the total of evaluable patients without residual disease after the first induction cycle with chemotherapy plus daratumumab

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Chiaretti, Principal Investigator — University of Roma La Sapienza
Locations (3):
- Italy (3):
  - Ematologia AOU Careggi, Florence
  - Ematologia P.O. Vito Fazzi - Lecce, Lecce
  - Ematologia AOU Policlinico Umberto I, Roma

IPD SHARING:
Plan to Share IPD: No